CLINICAL TRIAL: NCT03833570
Title: The Effectiveness of Melatonin in Prevention of Radiation-induced Oral Mucositis
Brief Title: Melatonin for Prevention of Radiation Induced Oral Mucositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Instructor of Dental Public Health, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0008839
Record Dates: First submitted 2019-02-03; First posted 2019-02-07 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Oral Mucositis (Ulcerative) Due to Radiation
Keywords: Melatonin
MeSH Terms: conditions — Stomatitis; Ulcer | interventions — Melatonin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Melatonin therapy (Experimental): Rapid Release Capsules Melatonin, 10 mg in combination with the symptomatic treatment
  Symptomatic treatment which included:
  * Miconaz oral gel
  * BBC oral spray
  * Oracure gel
  * Alkamisr sachets
  Melatonin capsules dose: Two tablets,30 minutes before sleeping once daily for six weeks
  Symptomatic treatment dose: Three times a day for six weeks
  Interventions: Dietary Supplement: Rapid Release Capsules Melatonin, 10 mg; Drug: Miconaz oral gel; Drug: BBC oral spray; Drug: Oracure gel; Other: Alkamisr sachets
- Conventional therapy (Active Comparator): Conventional therapy (symptomatic treatment) which included:
  * Miconaz oral gel
  * BBC oral spray
  * Oracure gel
  * Alkamisr sachets
  Dose: Three times a day for six weeks
  Interventions: Drug: Miconaz oral gel; Drug: BBC oral spray; Drug: Oracure gel; Other: Alkamisr sachets

INTERVENTIONS:
Dietary Supplement: Rapid Release Capsules Melatonin, 10 mg — Melatonin is a dietary supplement which is naturally produced in the body and closely involved in the natural sleep cycle. recently topical and systemic melatonin supplements. have been proposed as a new therapeutic modality for oral mucositis due to its anti-cancer, anti-inflammatory, and anti-oxidant effects.
  Arms: Melatonin therapy
Drug: Miconaz oral gel — Antifungal agent
Drug: BBC oral spray — Topical anesthetics and anti-inflammatory agent
Drug: Oracure gel — Topical analgesic gel
Other: Alkamisr sachets — Sodium bicarbonate mouthwash

SUMMARY:
The main aim of this study was to evaluate the effectiveness of melatonin in prevention of radiation induced oral mucositis clinically and biochemically.

DETAILED DESCRIPTION:
The study was designed as randomized, controlled, clinical trial. patients who were undergoing chemoradiation were divided into two groups: Group I: was given conventional treatment. Group II: was given melatonin therapy in combination with the conventional treatment.

All patients were clinically evaluated at the start the radiotherapy, three weeks and six weeks later for pain and oral mucositis severity. in addition, the total antioxidant capacity of the melatonin was evaluated at the start of the radiotherapy and six weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are going to receive radiotherapy as a treatment of head and neck cancer either as postoperative (adjuvant) therapy or definitive therapy.
* Patients whose radiotherapy treatment planned dose is between 60-70 Gy.
* Patients who had received chemotherapy prior to radiotherapy or are going to receive chemotherapy in concomitant to radiotherapy.

Exclusion Criteria:

* Patients under Anticoagulants such as warfarin, heparin, or aspirin.
* Patients under Fluvoxamine (Luvox) and Nifedipine medications.
* Patients whose radiotherapy treatment planned dose is lower than 60 Gy.
* Pregnant and lactating women.
* Patients suffering from any uncontrolled systemic diseases (such as diabetes, cardiovascular, liver disorder, renal dysfunction)
* Patients with findings of any physical or mental abnormality which would interfere with or be affected by the study procedure.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in severity of oral mucositis at different time points along the study | up to 3 and 6 weeks
  Oral mucositis will be evaluated by the World Health Organization (WHO) scale which record the extent and severity of oral mucositis at the third and sixth week after the first radiotherapy session.
  This scale combines both subjective and objective measures of oral mucositis.
  World Health Organization (WHO) scale for oral mucositis:
  * Grade 0 = No oral mucositis
  * Grade 1 = Erythema and Soreness
  * Grade 2 = Ulcers, able to eat solids
  * Grade 3 = Ulcers, requires liquid diet (due to mucositis)
  * Grade 4 = Ulcers, alimentation not possible (due to mucositis)
Changes in the total antioxidant capacity (TAC) in saliva at different time points along the study | Baseline (day 0) and up to 6 weeks
  TAC is an index that measures total capacity of antioxidants in biological fluids using Colorimetric Method. it can evaluate the antioxidant response against the free radicals produced by radiotherapy.
  Normal reference values for TAC in saliva: 0.3-1 mM/L Higher values than normal range indicate higher level of TAC
  Changes in the total antioxidant capacity were evaluated at the first day of radiotherapy session (baseline) and six weeks later

SECONDARY OUTCOMES:
Pain and discomfort severity at different time points along the study: Numeric Rating Scale | up to 3 and 6 weeks
  Discomfort and pain severity were reported by each patient using Numeric Rating Scale (NRS) at the third and sixth week after the first radiotherapy session.
  The NRS was calibrated from 0 to 10 with ranges tagged as;
  * No pain (NRS 0)
  * Mild pain (NRS 1-3)
  * Moderate pain (NRS 4-7)
  * Unbearable pain (NRS 8-10)

CONTACTS AND LOCATIONS:
Overall Officials: Hossam H Abdelaziz Elsabbagh, BDS, Principal Investigator — Alexandria University; Eglal M Moussa, Phd, Study Director — Alexandria University; Sabah AH Mahmoud, Phd, Study Director — University of Alexandria; Rasha O Elsaka, Phd, Study Director — University of Alexandria
Locations (1):
- Outpatient clinic of Department of Clinical Oncology, Faculty of Medicine, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feller L, Essop R, Wood NH, Khammissa RA, Chikte UM, Meyerov R, Lemmer J. Chemotherapy- and radiotherapy-induced oral mucositis: pathobiology, epidemiology and management. SADJ. 2010 Sep;65(8):372-4. PMID 21133051
- [Background] Duncan GG, Epstein JB, Tu D, El Sayed S, Bezjak A, Ottaway J, Pater J; National Cancer Institute of Canada Clinical Trials Group. Quality of life, mucositis, and xerostomia from radiotherapy for head and neck cancers: a report from the NCIC CTG HN2 randomized trial of an antimicrobial lozenge to prevent mucositis. Head Neck. 2005 May;27(5):421-8. doi: 10.1002/hed.20162. PMID 15782422
- [Background] Campos MI, Campos CN, Aarestrup FM, Aarestrup BJ. Oral mucositis in cancer treatment: Natural history, prevention and treatment. Mol Clin Oncol. 2014 May;2(3):337-340. doi: 10.3892/mco.2014.253. Epub 2014 Feb 7. PMID 24772297
- [Background] Harris DJ. Cancer treatment-induced mucositis pain: strategies for assessment and management. Ther Clin Risk Manag. 2006 Sep;2(3):251-8. doi: 10.2147/tcrm.2006.2.3.251. PMID 18360600
- [Background] Maria OM, Eliopoulos N, Muanza T. Radiation-Induced Oral Mucositis. Front Oncol. 2017 May 22;7:89. doi: 10.3389/fonc.2017.00089. eCollection 2017. PMID 28589080
- [Background] Sonis ST. Oral mucositis in cancer therapy. J Support Oncol. 2004 Nov-Dec;2(6 Suppl 3):3-8. PMID 15605918
- [Background] Lee CS, Ryan EJ, Doherty GA. Gastro-intestinal toxicity of chemotherapeutics in colorectal cancer: the role of inflammation. World J Gastroenterol. 2014 Apr 14;20(14):3751-61. doi: 10.3748/wjg.v20.i14.3751. PMID 24744571
- [Background] Villa A, Sonis ST. Mucositis: pathobiology and management. Curr Opin Oncol. 2015 May;27(3):159-64. doi: 10.1097/CCO.0000000000000180. PMID 25774860
- [Background] Volpato LE, Silva TC, Oliveira TM, Sakai VT, Machado MA. Radiation therapy and chemotherapy-induced oral mucositis. Braz J Otorhinolaryngol. 2007 Jul-Aug;73(4):562-8. doi: 10.1016/s1808-8694(15)30110-5. PMID 17923929
- [Background] Moslehi A, Taghizadeh-Ghehi M, Gholami K, Hadjibabaie M, Jahangard-Rafsanjani Z, Sarayani A, Javadi M, Esfandbod M, Ghavamzadeh A. N-acetyl cysteine for prevention of oral mucositis in hematopoietic SCT: a double-blind, randomized, placebo-controlled trial. Bone Marrow Transplant. 2014 Jun;49(6):818-23. doi: 10.1038/bmt.2014.34. Epub 2014 Mar 10. PMID 24614837
- [Background] Hardeland R, Pandi-Perumal SR, Cardinali DP. Melatonin. Int J Biochem Cell Biol. 2006 Mar;38(3):313-6. doi: 10.1016/j.biocel.2005.08.020. Epub 2005 Sep 27. PMID 16219483
- [Background] Brasure M, MacDonald R, Fuchs E, Olson CM, Carlyle M, Diem S, Koffel E, Khawaja IS, Ouellette J, Butler M, Kane RL, Wilt TJ. Management of Insomnia Disorder [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2015 Dec. Report No.: 15(16)-EHC027-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK343503/ PMID 26844312
- [Background] Lyseng-Williamson KA. Melatonin prolonged release: in the treatment of insomnia in patients aged >/=55 years. Drugs Aging. 2012 Nov;29(11):911-23. doi: 10.1007/s40266-012-0018-z. PMID 23044640
- [Background] Lemoine P, Zisapel N. Prolonged-release formulation of melatonin (Circadin) for the treatment of insomnia. Expert Opin Pharmacother. 2012 Apr;13(6):895-905. doi: 10.1517/14656566.2012.667076. Epub 2012 Mar 19. PMID 22429105
- [Background] Zisapel N. [Controlled release melatonin (Circadin) in the treatment of insomnia in older patients: efficacy and safety in patients with history of use and non-use of hypnotic drugs]. Harefuah. 2009 May;148(5):337-41, 348. Hebrew. PMID 19630367
- [Background] Zhang HM, Zhang Y. Melatonin: a well-documented antioxidant with conditional pro-oxidant actions. J Pineal Res. 2014 Sep;57(2):131-46. doi: 10.1111/jpi.12162. Epub 2014 Aug 6. PMID 25060102
- [Background] Najeeb S, Khurshid Z, Zohaib S, Zafar MS. Therapeutic potential of melatonin in oral medicine and periodontology. Kaohsiung J Med Sci. 2016 Aug;32(8):391-6. doi: 10.1016/j.kjms.2016.06.005. Epub 2016 Jul 25. PMID 27523451
- [Background] Wang YM, Jin BZ, Ai F, Duan CH, Lu YZ, Dong TF, Fu QL. The efficacy and safety of melatonin in concurrent chemotherapy or radiotherapy for solid tumors: a meta-analysis of randomized controlled trials. Cancer Chemother Pharmacol. 2012 May;69(5):1213-20. doi: 10.1007/s00280-012-1828-8. Epub 2012 Jan 24. PMID 22271210
- [Background] McCormack HM, Horne DJ, Sheather S. Clinical applications of visual analogue scales: a critical review. Psychol Med. 1988 Nov;18(4):1007-19. doi: 10.1017/s0033291700009934. PMID 3078045
- [Background] Koracevic D, Koracevic G, Djordjevic V, Andrejevic S, Cosic V. Method for the measurement of antioxidant activity in human fluids. J Clin Pathol. 2001 May;54(5):356-61. doi: 10.1136/jcp.54.5.356. PMID 11328833
- [Background] Rai B, Kaur J, Jacobs R, Singh J. Possible action mechanism for curcumin in pre-cancerous lesions based on serum and salivary markers of oxidative stress. J Oral Sci. 2010 Jun;52(2):251-6. doi: 10.2334/josnusd.52.251. PMID 20587949
- [Background] Mihandoost E, Shirazi A, Mahdavi SR, Aliasgharzadeh A. Can melatonin help us in radiation oncology treatments? Biomed Res Int. 2014;2014:578137. doi: 10.1155/2014/578137. Epub 2014 May 11. PMID 24900972
- [Background] Shirzad A, Pouramir M, Seyedmajidi M, Jenabian N, Bijani A, Motallebnejad M. Salivary total antioxidant capacity and lipid peroxidation in patients with erosive oral lichen planus. J Dent Res Dent Clin Dent Prospects. 2014 Winter;8(1):35-9. doi: 10.5681/joddd.2014.006. Epub 2014 Mar 5. PMID 25024837
- See also: WHO Handbook for Reporting Results of Cancer Treatment — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2010938/